CLINICAL TRIAL: NCT03970824
Title: A Phase 1, Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of CT-P17 and Humira (US-licensed Humira and EU-approved Humira) in Healthy Subjects
Brief Title: To Compare the Pharmacokinetics and Safety of CT-P17 and Humira in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-P17 1.1
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — CT-P17

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CT-P17 (Experimental): a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P17
- US-licensed Humira (Active Comparator): a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: US-licensed Humira
- EU-approved Humira (Active Comparator): a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: EU-approved Humira

INTERVENTIONS:
Biological: CT-P17 — 40 mg/0.4ml (100 mg/mL) administered as a single SC injection via PFS
  Arms: CT-P17
Biological: US-licensed Humira — 40 mg/0.4ml (100 mg/mL) administered as a single SC injection via PFS
  Arms: US-licensed Humira
Biological: EU-approved Humira — 40 mg/0.4ml (100 mg/mL) administered as a single SC injection via PFS
  Arms: EU-approved Humira

SUMMARY:
This is a Phase 1, Randomized, Double-blind, Three-arm, Parallel group, Single-dose Study to Compare the Pharmacokinetics and Safety of CT-P17 and Humira (US licensed Humira and EU-approved Humira) in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* BMI between 18.0 and 29.9 kg/m2, both inclusive, when rounded to the nearest tenth

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or current infection of hepatitis B virus (except for past resolved infection), hepatitis C virus, human immunodeficiency virus, or syphilis
* Active or latent Tuberculosis
* History of malignancy
* Previous monoclonal antibody or fusion protein treatment, or current use of any biologic
* Planning to be pregnant or father a child or donate sperm within 5 month after administration
* Undergone treatment with an investigational drug or participated in another clinical trial within 90 days or 5 half-lives (whichever is longer)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 312 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Joon Lee, Study Director — Celltrion, Inc.
Locations (9):
- South Korea (9):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Busan Paik Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu KS, Jang IJ, Lim HS, Hong JH, Kim MG, Park MK, Cho DY, Park MS, Chung JY, Ghim JL, Lee S, Yoon SK, Kwon IS, Lee SJ, Kim SH, Bae YJ, Cha JB, Furst DE, Keystone E, Kay J. Pharmacokinetic equivalence of CT-P17 to high-concentration (100 mg/ml) reference adalimumab: A randomized phase I study in healthy subjects. Clin Transl Sci. 2021 Jul;14(4):1280-1291. doi: 10.1111/cts.12967. Epub 2021 Mar 2. PMID 33503313

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
Started | 103 | 103 | 106
Completed | 101 | 100 | 102
Not Completed | 2 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (all randomly assigned subjects who received a complete or partial dose of study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira | Total
Number analyzed (Participants) | 102 | 102 | 104 | 308
Age, Continuous [Median (Full Range); unit: years] | 25.0 [19 to 51] | 26.0 [19 to 53] | 26.0 [19 to 54] | 26.0 [19 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 15 | 44
  Male | 87 | 88 | 89 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 102 | 102 | 104 | 308
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 102 | 102 | 104 | 308
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 102 | 102 | 104 | 308

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf)
Description: Primary endpoints were equivalence of PK between CT-P17 and reference drugs in terms of AUC0-inf, AUC0-last, and Cmax. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.
Time Frame: up to Day 71
Population: Pharmacokinetic population (all randomly assigned subjects who received a complete dose of study drug and provided at least 1 post-treatment serum concentration above the lower limit of quantification for adalimumab)
Measure: Mean (Standard Deviation); unit: h•μg/mL
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
Number analyzed (Participants) | 80 | 86 | 89
h•μg/mL | 2656.5 (1150.16) | 2469.7 (917.47) | 2690.6 (943.76)
Statistical Analysis 1: Comparison: CT-P17 vs US-licensed Humira; Statistical analysis of primary PK parameters was performed using an analysis of covariance model (ANCOVA) including covariates for gender, study center, and body weight; Test type: Equivalence — PK equivalence was concluded if 90% confidence intervals (CIs) for percent ratios of geometric least squares means in AUC0-inf, AUC0-last, and Cmax were within the equivalence margin of 80-125%; Ratio of geometric least squares means = 105.79, 90% CI 2-sided [97.19 to 115.16]
Statistical Analysis 2: Comparison: US-licensed Humira vs EU-approved Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 92.63, 90% CI 2-sided [85.29 to 100.61]
Statistical Analysis 3: Comparison: CT-P17 vs EU-approved Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 98.00, 90% CI 2-sided [90.06 to 106.63]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last)
Description: as for outcome 1
Time Frame: up to Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h•μg/mL
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
Number analyzed (Participants) | 96 | 93 | 98
h•μg/mL | 2372.7 (954.82) | 2185.0 (795.91) | 2394.7 (866.95)
Statistical Analysis 1: Comparison: CT-P17 vs US-licensed Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 107.30, 90% CI 2-sided [98.29 to 117.13]
Statistical Analysis 2: Comparison: US-licensed Humira vs EU-approved Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 93.93, 90% CI 2-sided [86.08 to 102.50]
Statistical Analysis 3: Comparison: CT-P17 vs EU-approved Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 100.79, 90% CI 2-sided [92.42 to 109.92]

3. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: as for outcome 1
Time Frame: up to Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
Number analyzed (Participants) | 96 | 93 | 98
μg/mL | 3.619 (1.3522) | 3.556 (1.1972) | 3.660 (1.2212)
Statistical Analysis 1: Comparison: CT-P17 vs US-licensed Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 101.89, 90% CI 2-sided [95.33 to 108.89]
Statistical Analysis 2: Comparison: US-licensed Humira vs EU-approved Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 98.20, 90% CI 2-sided [91.91 to 104.92]
Statistical Analysis 3: Comparison: CT-P17 vs EU-approved Humira; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of geometric least squares means = 100.05, 90% CI 2-sided [93.69 to 106.85]

4. Secondary Outcome: Time to the Maximum Serum Concentration (Tmax)
Description: The secondary objective was to evaluate the additional PK parameters including Tmax and t1/2. Blood samples for PK analysis were obtained pre-dose and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504, 672, 1008, 1344, and 1680 hour post-dose.
Time Frame: up to Day 71
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
Number analyzed (Participants) | 96 | 93 | 98
h | 167.433 [48.00 to 504.08] | 166.833 [48.00 to 433.22] | 144.000 [48.00 to 671.35]

5. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: as for outcome 4
Time Frame: up to Day 71
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
Number analyzed (Participants) | 80 | 86 | 89
h | 340.3 (163.61) | 331.3 (165.05) | 339.5 (151.04)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time the ICF was signed and until the end of the subject's participation in the study (up to Day 71).
Description: Only treatment-emergent adverse events and treatment-emergent serious adverse events were summarized.
Arm/Group | CT-P17 | US-licensed Humira | EU-approved Humira
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 2/102 | 0/102 | 1/104
Other Adverse Events (participants affected / at risk) | 26/102 | 27/102 | 27/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P17 (N=102) | US-licensed Humira (N=102) | EU-approved Humira (N=104)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P17 (N=102) | US-licensed Humira (N=102) | EU-approved Humira (N=104)
Injection site reaction (General disorders) | 20 | 16 | 19
Nasopharyngitis (Infections and infestations) | 3 | 7 | 3
Headache (Nervous system disorders) | 6 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT03970824/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03970824/SAP_001.pdf